CLINICAL TRIAL: NCT05924139
Title: Omega-3 Fatty Acid Supplementation to Enhance Performance in Collegiate Athletes
Brief Title: Omega-3 Fatty Acid Supplementation to Enhance Performance
Acronym: FO n-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1994931
Record Dates: First submitted 2023-06-05; First posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Strength; Body Composition; Muscle Soreness
Keywords: omega-3 fatty acid; strength; body composition; muscle soreness
MeSH Terms: conditions — Myalgia | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega-3 fatty acid (Experimental): Nordic Naturals (Ultimate Omega) will be used as the intervention at a dose of 4 grams/day (3840 mg total fish oil with 1950 mg EPA and 1350 mg DHA
  Interventions: Dietary Supplement: Omega-3 fatty acid
- Coconut oil (Placebo Comparator): dose of 4 grams/day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 fatty acid — 6 capsules per day of 3840 mg that included 1950 mg EPA and 1350 mg DHA
  Other Names: Nordic Naturals Ultimate Omega
  Arms: Omega-3 fatty acid
Dietary Supplement: Placebo — 4 capsules per day of coconut oil
  Arms: Coconut oil

SUMMARY:
The goal of this intervention study is to determine if omega-3 fatty acid supplementation as compared to placebo improves performance in track and field athletes. The main questions it aims to answer are:

1. Can performance be improved
2. Can strength be enhanced
3. Will positive body composition changes occur (lean vs fat mass)
4. Will feelings of muscle soreness be diminished Participants will take either omega-3 fatty acid supplements or placebo and continue with their sport specific training regimen.

Researchers will compare the supplement group to placebo group to determine if there are any significant differences.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled trial to determine the efficacy of fish oil-derived omega-3 fatty acid supplementation. Up to sixty participants will be randomized to receive one of two conditions: 4.0 grams of FO n-3/day or placebo (coconut oil) for the 10-week protocol study period. Nordic Naturals (Ultimate Omega) will be used as the intervention at a dose of 6 capsules/day (3840 mg total FO/1950 mg EPA/1350 mg DHA). Although protocols have varied among studies with regards to dosage, the proposed regimen was selected based on studies on strength in older adults and college-aged athletes utilizing a range of 2-5g FO n-3 per day. Blinded randomization will be accomplished with a research associate providing every first (of two) participants the placebo, while the second will receive the supplemented condition until recruitment is complete. Participants will be provided their supplement in 2-week increments and instructed to consume with/near their evening meal. Used bottles will be returned after two weeks and participants will receive the next 2-week supply of supplement and the leftover pill count will determine compliance rate.

The target population is apparently healthy college athletes (male and female of all ethnicities) between the ages of 18-25 years at Baylor University. Participants must be able to read and understand English and sign their own consent form. Up to 60 subjects will be recruited via direct contact or team briefings with permission of the coaches.

ELIGIBILITY:
Inclusion Criteria:

Apparently healthy college athletes (male and female of all ethnicities) between the ages of 18-25 years.

Exclusion Criteria: -Participants will be excluded if they are unable to physically train due to injury/illness or are pregnant, or have a known heart condition or pacemaker.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Strength | change from baseline at 8 weeks
  lower body strength will be evaluated via a counter movement jump
Power | change from baseline at 8 weeks
  handgrip strength will be used as a proxy for upper body strength via a dynamometer

SECONDARY OUTCOMES:
Body composition | change from baseline at 8 weeks
  bioelectrical impedance analysis (BIA), a double-indirect body composition technique based on a 3-component model (fat mass, fat-free mass, and total body water), will be performed.
Muscle soreness | change from baseline, every 2 weeks and at 8 weeks
  Subjects will be asked to rate their muscle soreness on a 10-point Likert scale
Omega-3 index | change from baseline at 8 weeks
  The Omega-3 Index provides information on the participants baseline level of EPA/DHA level in the blood

CONTACTS AND LOCATIONS:
Overall Officials: LesLee Funderburk, Principal Investigator — Associate professor
Locations (1):
- Baylor University, Waco, Texas, United States

IPD SHARING:
Plan to Share IPD: No